CLINICAL TRIAL: NCT00002393
Title: A Phase III, Double-Blind, Placebo-Controlled, Multicenter Study to Determine the Effectiveness and Tolerability of the Combination of DMP 266 and Indinavir Versus Indinavir in HIV-Infected Patients Receiving Nucleoside Analogue (NRTI) Therapy
Brief Title: A Study of Indinavir Taken With or Without DMP 266
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dupont Merck (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 281A; DMP 266-020
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-07

CONDITIONS: HIV Infections
Keywords: Placebos; Drug Therapy, Combination; HIV Protease Inhibitors; Indinavir; Reverse Transcriptase Inhibitors; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; efavirenz

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Efavirenz

SUMMARY:
The purpose of this study is to see if it is safe and effective to add DMP 266 to an anti-HIV treatment program of indinavir and nucleoside reverse transcriptase inhibitors (NRTIs).

DETAILED DESCRIPTION:
In this double-blind, placebo-controlled study, 300 patients are randomized to 1 or 2 reverse transcriptase inhibitors of their choice plus blinded therapy on Arm A or B as follows:

Arm A: DMP 266 placebo plus indinavir. Arm B: DMP 266 plus indinavir. After 16 weeks, patients may switch the NRTI portion of their regimen if they meet a treatment failure criterion. After the completion of the 24-week period, patients have the option to continue on open-label DMP 266 and indinavir.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* CD4+ cell count of at least 50 cells/mm3.
* HIV RNA level of at least 10,000 copies/ml by reverse transcriptase polymerase chain reaction (RT-PCR, Amplicor test kit) at screening.
* Signed, informed consent from parent or legal guardian for patients less than 18 years of age.

Exclusion Criteria

Prior Medication:

Excluded:

* DMP 266.
* Other nonnucleoside reverse transcriptase inhibitors.

Required:

One or two NRTIs (except ZDV and d4T in combination) for a minimum of 8 weeks, within 12 weeks prior to screening.

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300

CONTACTS AND LOCATIONS:
Locations (12):
- United States (9):
  - Kaiser Foundation Hospital, San Francisco, California
  - Med College of Georgia, Augusta, Georgia
  - Chicago Ctr for Clinical Research, Chicago, Illinois
  - Univ of Kentucky Med Ctr / Chandler Med Ctr, Lexington, Kentucky
  - Tulane Univ / Tulane / LSU Clinical Trials Unit, New Orleans, Louisiana
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - Vanderbilt Univ, Nashville, Tennessee
  - Hampton Roads Med Specialists, Hampton, Virginia
- Canada (2):
  - Southern Alberta HIV Clinic / Foot Hills Hosp, Calgary, Alberta
  - Ottawa Gen Hosp, Ottawa, Ontario
- Univ of Puerto Rico School of Medicine, San Juan, Puerto Rico

REFERENCES:
- [Background] Haas DW, Fessel WJ, Delapenha RA, Kessler H, Seekins D, Kaplan M, Ruiz NM, Ploughman LM, Labriola DF, Manion DJ. Therapy with efavirenz plus indinavir in patients with extensive prior nucleoside reverse-transcriptase inhibitor experience: a randomized, double-blind, placebo-controlled trial. J Infect Dis. 2001 Feb 1;183(3):392-400. doi: 10.1086/318083. Epub 2000 Dec 29. PMID 11133370